CLINICAL TRIAL: NCT04960215
Title: Coenzyme Q10 as Treatment for Long Term COVID-19
Acronym: QVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Pharma Nord (Industry)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QVID-001
Record Dates: First submitted 2021-06-11; First posted 2021-07-13 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2021-06

CONDITIONS: Covid19; Long Term Covid19
Keywords: Coenzyme Q10
MeSH Terms: conditions — COVID-19 | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 (Active Comparator)
  Interventions: Drug: Coenzyme Q10
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Coenzyme Q10 — Coenzyme Q10 (myoquinon) capsule 100mg, 5 capsules a day.
  Other Names: Myoquinon
  Arms: Coenzyme Q10
Drug: Placebo — A soft gelatin capsule containing soy oil, 5 capsules a day.
  Arms: Placebo

SUMMARY:
This study is a randomized, placebo-controlled, double-blinded, cross-over designed clinical trial investigating the effect of high-dose Coenzyme Q10 treatment in subjects with persisting symptoms more than 12 weeks af SARS-CoV-2 infection, Long Term COVID-19 (LTC).

DETAILED DESCRIPTION:
The aim is to investigate the effect of high-dose Coenzyme Q10 on number and severity of self-reported symptoms in patients with Long Term COVID-19.

The study will be conducted at the Department of Infectious Diseases, Aarhus University Hospital in the LTC Outpatient Clinic. 120 study participants will be randomized 1:1 to receive placebo or CoQ10 in a dose of 500mg/day for 6 weeks. After a wash-out period of 4 weeks, participants are allocated to the opposite treatment for 6 weeks. The EQ-5D-5L and an LTC-specific questionnaire are completed at baseline and after 6,10,16, and 20 weeks. At each of 5 visits blood samples will be collected from the participants for immunological investigations and assessment of cellular metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Able to give informed consent.
* History of documented SARS-CoV-2 infection either by RT-PCR or antibody test.
* Symptoms related to Long Term COVID-19, defined as being investigated, diagnosed and followed by specialized infectious diseases physicians in the Long Term COVID-19 Outpatient Clinic, Central Region of Denmark, Aarhus University Hospital.
* Symptoms not attributable to other co-morbidity/condition.

Exclusion Criteria:

* Symptoms of acute COVID-19, as defined by The Danish Health Authorities.
* Women who are pregnant or breastfeeding, or with a positive pregnancy test as determined by a positive urine beta-human chorionic gonadotropin test during screening
* Hypersensitivity to the active ingredient or to any excipient of the medicinal product
* Known allergy to soy or peanuts.
* Individuals with reduced kidney or liver-function.
* Patients in anticoagulant therapy with vitamin K antagonists.
* Any condition that, in the Investigator's opinion, will prevent adequate compliance with study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Effect of Coenzyme Q10 treatment in Long Term COVID-19 on number of self-reported symptoms of LTC measured by EQ-5D-5L questionnaire. | Changes from baseline questionnaire response to questionnaire response after 6 weeks of treatment
  Number of self-reported symptoms measured by EQ-5D-5L questionnaire.
Effect of Coenzyme Q10 treatment in Long Term COVID-19 on number of self-reported symptoms of LTC measured by Long Term COVID-specific questionnaire. | Changes from baseline questionnaire response to questionnaire response after 6 weeks of treatment
  Number of self-reported symptoms measured by Long Term COVID-specific questionnaire.
Effect of Coenzyme Q10 treatment in Long Term COVID-19 on severity (symptoms score) of self-reported symptoms of LTC measured by Long Term COVID-specific questionnaire. | Changes from baseline questionnaire response to questionnaire response after 6 weeks of treatment
  Severity by symptom score of self-reported symptoms measured by Long Term COVID-specific questionnaire. The questionnaire consist of 32 questions with a graduation of 0-4, thus maximum number of points is 128 implying a high number of severe symptoms.
Effect of Coenzyme Q10 treatment in Long Term COVID-19 on severity (symptoms score) of self-reported symptoms of LTC measured by EQ-5D-5L questionnaire. | Changes from baseline questionnaire response to questionnaire response after 6 weeks of treatment
  Severity by symptom score of self-reported symptoms measured by ED-5Q-5L questionnaire. The questionnaire consist of 5 questions with a graduation of 0-4, thus maximum number of points is 20 implying a high number of severe symptoms.

SECONDARY OUTCOMES:
Prolonged effect of Coenzyme Q10 treatment in Long Term COVID-19 on number of self-reported symptoms of LTC measured by Long Term COVID-specific questionnaire. | Changes from baseline questionnaire response to questionnaire response 4 weeks after ended treatment.
  Number of self-reported symptoms measured by Long Term COVID-specific questionnaire.
Prolonged effect of Coenzyme Q10 treatment in Long Term COVID-19 on number of self-reported symptoms of LTC measured by EQ-5D-5L questionnaire. | Changes from baseline questionnaire response to questionnaire response 4 weeks after ended treatment.
  Number of self-reported symptoms measured by EQ-5D-5L questionnaire.
Prolonged effect of Coenzyme Q10 treatment in Long Term COVID-19 on severity (symptoms score) of self-reported symptoms of LTC measured by Long Term COVID-specific questionnaire. | Changes from baseline questionnaire response to questionnaire response 4 weeks after ended treatment.
  Severity by symptom score of self-reported symptoms measured by Long Term COVID-specific questionnaire. The questionnaire consist of 32 questions with a graduation of 0-4, thus maximum number of points is 128 implying a high number of severe symptoms.
Prolonged effect of Coenzyme Q10 treatment in Long Term COVID-19 on severity (symptoms score) of self-reported symptoms of LTC measured by EQ-5D-5L questionnaire. | Changes from baseline questionnaire response to questionnaire response 4 weeks after ended treatment.
  Severity by symptom score of self-reported symptoms measured by ED-5Q-5L questionnaire. The questionnaire consist of 5 questions with a graduation of 0-4, thus maximum number of points is 20 implying a high number of severe symptoms.
Safety and tolerability of treatment with high-dose Coenzyme Q10 as measured by number of adverse events, adverse reactions, serious adverse events and serious adverse reactions. | End of data collection after 20 weeks.
  Safety evaluation by incidence of adverse events, adverse reactions, serious adverse events and serious adverse reactions.

OTHER OUTCOMES:
Presence of auto-reactive antibodies in Long Term COVID-19 | Blood samples week 6, 10, 16 and 20 after enrollment
  Investigation of auto-reactive antibodies at baseline compared to healthy controls (biobank samples), by immunohistochemistry and enzyme-linked immunosorbent assay (ELISA) against tissue proteins.
Assessment of levels of Coenzyme Q10 plasma and PBMC in Long Term COVID-19 patients treated with Coenzyme Q10 versus placebo. | Blood samples after 6 weeks of treatment and after 6 weeks of placebo.
  Assessment of baseline levels Coenzyme Q10 in plasma (nmol/L) and in PBMC (picogram / mg protein) , measured by High Performance Liquid Chromatography (HPLC), as this parameter previously has been associated with fatigue.
Quantitative proteomics in peripheral blood mononuclear cells (PBMCs) from Coenzyme Q10 treated patients versus placebo. | Blood samples week 6, 10, 16 and 20 after enrollment
  Relative quantification of the approximately four thousand most abundant proteins is performed by liquid chromatography (LC) tandem mass spectrometry (MS/MS). The quantitative signal is the MS peak intensities, with arbitrary scale. Statistically differentially regulated proteins are filtered out and described specifically.
Assessment of cellular metabolic activity in PBMCs from Coenzyme Q10 treated patients by Seahorse analysis versus placebo. | Blood samples week 6, 10, 16 and 20 after enrollment
  Differential analysis of metabolic activities (Seahorse) in PBMCs from the treated patients versus placebo. Extracellular Acidification Rate (ECAR) (picomoles protons / minute) and Oxygen Consumption Rate (OCR) (picomoles O2 per minute) are measured to estimate glycolytic rate and respiration rates in the isolated PBMCs, respectively.
Analysis of oxidative stress marker 8-isoprostane in Long Term COVID-19 patients treated with Coenzyme Q10 versus placebo. | Blood samples week 6, 10, 16 and 20 after enrollment
  Differential analysis of plasma samples from CoQ10 treated patients versus placebo, with respect to the oxidative stress marker 8-isoprostane by ELISA assay measured in picomoles 8-isoprostane per mL.
Assessment of presence of cytokines in Long Term COVID-19 patients treated with Coenzyme Q10 versus placebo. | Blood samples week 6, 10, 16 and 20 after enrollment
  Differential analysis of plasma samples from CoQ10 treated patients versus placebo with Luminex to assess presence of cytokines measured as picomole cytokine / mL.
Analysis of metabolites of the kynurenic pathway in Long Term COVID-19 patients treated with Coenzyme Q10 versus placebo. | Blood samples week 6, 10, 16 and 20 after enrollment
  Differential analysis of plasma samples from CoQ10 treated patients versus placebo with respect to metabolites of the kynurenic pathway by LC-MS/MS measured in nanomole per mL.

CONTACTS AND LOCATIONS:
Overall Officials: Line Khalidan Vibholm, M.D., Ph.D, Principal Investigator — Department of Infections Diseases, Aarhus University Hospital
Locations (1):
- Department of Infectious Diseases, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hansen KS, Mogensen TH, Agergaard J, Schiottz-Christensen B, Ostergaard L, Vibholm LK, Leth S. High-dose coenzyme Q10 therapy versus placebo in patients with post COVID-19 condition: a randomized, phase 2, crossover trial. Lancet Reg Health Eur. 2023 Jan;24:100539. doi: 10.1016/j.lanepe.2022.100539. Epub 2022 Nov 2. PMID 36337437